CLINICAL TRIAL: NCT06311656
Title: A Placebo-controlled, Phase 1, Participant- and Investigator-blinded, Single- and Multiple- Dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of LY4100511 (DC-853) in Healthy Asian and Non-Asian Participants
Brief Title: A Study to Evaluate Safety, Tolerability of LY4100511 (DC-853) in Healthy Asian and Non-Asian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DICE Therapeutics, Inc., a wholly owned subsidiary of Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 18840; J5C-MC-FOAA (Other: DICE Therapeutics, a wholly owned subsidiary of Eli Lilly and Company); DCE853107 (Other: DICE Therapeutics, a wholly owned subsidiary of Eli Lilly and Company)
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- LY4100511 (DC-853) Part A Fasted (Experimental): Single and multiple doses of LY4100511 (DC-853) administered orally.
  Interventions: Drug: LY4100511 (DC-853)
- LY4100511 (DC-853) Part B (Experimental): Single and multiple higher doses of LY4100511 (DC-853) administered orally.
  Interventions: Drug: LY4100511 (DC-853)
- LY4100511 (DC-853) Part C (Open Label) (Experimental): Single dose of LY4100511 (DC-853) administered orally in fed and fasted states.
  Interventions: Drug: LY4100511 (DC-853)
- LY4100511 (DC-853) Part D (Experimental): Multiple higher doses of LY4100511 (DC-853) administered orally.
  Interventions: Drug: LY4100511 (DC-853)
- Placebo (Placebo Comparator): Placebo administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY4100511 (DC-853) — Administered orally fasted
  Arms: LY4100511 (DC-853) Part A Fasted
Drug: LY4100511 (DC-853) — Administered orally fasted.
  Arms: LY4100511 (DC-853) Part B
Drug: LY4100511 (DC-853) — Administered orally fed and fasted.
  Arms: LY4100511 (DC-853) Part C (Open Label)
Drug: LY4100511 (DC-853) — Administered orally fed and fasted.
  Arms: LY4100511 (DC-853) Part D
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess the safety and tolerability of LY4100511 (DC-853) after single and multiple dose administrations in healthy asian participants and non-Asian participants. Part A consists of 2 groups and Part B, C, and D include optional groups.

DETAILED DESCRIPTION:
Part B and C added per protocol amendment (May 2024) Added Part B to explore higher dose levels and Part C to explore effects of food. Part D added per protocol amendment (June 2024) to explore higher multiple doses.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are overtly healthy as determined by medical history, vital signs, and physical examination.
* Participants of Japanese, Chinese, and Non-Asian ethnicities
* Have a body mass index within the range of 18.0 to 32 kilograms per square meter (kg/m²). For healthy Japanese participants, have a body mass index of 18.0 to 28.0 kg/m²
* Have venous access sufficient to allow for blood sampling
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures

Exclusion Criteria:

* Have a current or recent acute, active infection
* Had any surgical procedure within 12 weeks prior to study
* Are immunocompromised
* Have presence of significant uncontrolled cerebro-cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, neurologic or neuropsychiatric disorders or abnormal laboratory values
* Are currently enrolled in a clinical study involving any experimental antibody or biologic therapy within the previous 6 months, or any other experimental therapy within 30 days before the first dose of the study intervention or during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with one or more Treatment Emergent Adverse Event(s) (TEAEs) and Serious Adverse Event(s) (SAEs) | Baseline up to 47 days
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module.

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY4100511 (DC-853) | Predose up to 47 days
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY4100511 (DC-853) | Predose up to 47 days

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Altasciences Clinical Los Angeles, Inc, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No